CLINICAL TRIAL: NCT06789302
Title: A Double-Blind, Randomized, Placebo-Controlled Phase IIa Clinical Trial to Evaluate the Safety and Efficacy of DT2-SCT in Subjects With Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Global Institute of Stem Cell Therapy and Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIOSTAR-001-2024
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: DT2-SCT Infusion (Experimental): Group A will be given DT2-SCT suspended on Plasma-Lyte A.
  Interventions: Drug: DT2-SCT intravenous infusion
- Group B: Placebo Treatment (Placebo Comparator): Group B will be given Plasma-Lite A only.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DT2-SCT intravenous infusion — DT2-SCT is an investigational therapy using autologous adipose-derived mesenchymal stem cells (MSCs) prepared from each participant's adipose tissue. MSCs are isolated from approximately 50 mL of adipose tissue obtained through a tumescent liposuction procedure. The cells are expanded, tested for contaminants, and suspended in a sterile, cryopreservation-free medium (Plasma-Lyte A) for administration.
  The intervention involves a single intravenous infusion of DT2-SCT at a dosage of 1 x 10^6 MSCs/kg body weight, delivered over a period of one hour. Participants will be closely monitored for at least two hours post-infusion to assess immediate safety and potential adverse effects.
  Arms: Group A: DT2-SCT Infusion
Other: Placebo — Participants in the placebo group (Group B) will receive a single intravenous infusion of Plasma-Lyte A, a sterile, isotonic, non-pyrogenic crystalloid solution. The infusion will be administered in a volume of 100 mL over a period of one hour.
  Arms: Group B: Placebo Treatment

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of DT2-SCT, a therapy using autologous adipose-derived mesenchymal stem cells, in adults with Type 2 Diabetes Mellitus (T2DM). The study aims to determine if DT2-SCT can reduce insulin resistance, improve blood sugar levels, and decrease the need for insulin or oral glucose-lowering medications.

Participants will be randomly assigned to receive either DT2-SCT or a placebo. They will undergo a single intravenous infusion after a liposuction procedure to collect adipose tissue, which will be processed to isolate stem cells for the therapy.

The study involves follow-up visits over six months to monitor safety, insulin resistance, blood sugar control, and any potential side effects.

DETAILED DESCRIPTION:
This clinical trial is a double-blind, randomized, placebo-controlled Phase IIa study to evaluate the safety and efficacy of DT2-SCT, an autologous adipose-derived mesenchymal stem cell (MSC) therapy, in adults with Type 2 Diabetes Mellitus (T2DM). The study will explore the potential of DT2-SCT to improve glycemic control, reduce insulin resistance, and decrease dependency on insulin and oral glucose-lowering drugs.

Study Design:

The trial involves 120 participants, randomized in a 1:1 ratio to receive either DT2-SCT or a placebo. The investigational product, DT2-SCT, consists of MSCs isolated from each participant's adipose tissue obtained via a tumescent liposuction procedure. The cells are processed, expanded, and prepared in a sterile, cryopreservation-free medium for a single intravenous infusion. The placebo consists of Plasma-Lyte A without MSCs.

Intervention and Monitoring:

Participants will undergo:

Screening and Enrollment: Eligibility will be determined based on inclusion and exclusion criteria, including a comprehensive review of medical history, laboratory tests, and diabetes status.

Liposuction Procedure: Approximately 50 mL of adipose tissue will be collected from the lower abdominal region under local anesthesia. The extracted tissue will be processed to isolate and expand MSCs.

Infusion Phase: Participants will receive either DT2-SCT (1 x 10^6 cells/kg) or placebo in a 100 mL Plasma-Lyte solution via intravenous infusion over one hour. Safety will be monitored during and after the infusion.

Follow-Up Visits: Participants will be followed for six months, with evaluations at 7 days, 1 month, 3 months, and 6 months post-infusion. These visits include assessments of glycemic control, insulin resistance, adverse events, and overall health.

Objectives:

Primary Objective: To determine the safety and tolerability of a single intravenous dose of DT2-SCT in T2DM patients.

Secondary Objectives:

Assess changes in insulin resistance using the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR).

Evaluate changes in fasting blood glucose (FBG) and HbA1c levels compared to baseline.

Measure the reduction in insulin and oral glucose-lowering drug dosages.

Methodology:

The MSCs used in DT2-SCT are self-renewing, multipotent cells with documented capacity for differentiation into various cell types, including pancreatic β-cells. The mechanism of action includes immunomodulation, anti-inflammatory effects, and potential enhancement of β-cell regeneration. These properties suggest that DT2-SCT could address both insulin resistance and β-cell dysfunction in T2DM.

Statistical Considerations:

The sample size of 120 participants is designed to provide robust safety data and meaningful descriptive results for efficacy. An interim safety analysis will be conducted after the first 20 participants complete their 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or female) between ages of 30 - 75 years
* Should have Type 2 diabetes mellitus
* With Insulin requirement of 0.7 IU/kg/d or 50 IU/d, whichever is lesser
* Glutamic acid decarboxylase (GAD) antibody status should be negative
* Body Mass Index (BMI) 19 - 30 kg/m2
* Fasting blood glucose (FBG) should be ≥ 7.0 mmol/L, and HbAc1 ≥ 7%
* Intravenous insulin tolerance tests (ITT) indicate a patient's insulin resistance
* Should be ambulatory and in good general health
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions
* Willing to abstain from the use of protocol-restricted treatments from Screening through the End-of-Treatment
* No clinically significant abnormalities observed in medical history, physical exam vital signs, and laboratory assessments
* For females with reproductive potential: Should agree to use effective contraception for at least 1 month prior to screening and should agree to use such a method till end of the study period and negative pregnancy test
* For males with reproductive potential: should use condoms and other methods to ensure effective contraception with a partner

Exclusion Criteria:

* Subjects with Type 1 Diabetes Mellitus (T1DM) or secondary diabetes
* Subjects with serum creatinine 1.5 mg/dl or higher
* Abnormal liver function test (defined as value of transaminases > 3 times the upper limit of normal or serum bilirubin higher than normal for the reference value for the laboratory)
* History of myocardial infarction or unstable angina in previous 3 months
* History of malignancy or current malignancy other than non-melanomatous skin cancer
* Subjects with active infections
* Subject with serious medical conditions other than cardiovascular disease
* Subject with, or with a medical history of auto-immune diseases
* Subject with a medical history of mental disorder or epilepsy
* Subject abuse alcohol 10 times a week or smoke 25 cigarettes a day
* Subject who was diagnosed with cancer within 5 years before screening
* Subject who participated in another clinical trial within 6 months prior to the screening of this clinical trial
* Subject who was administered with immunosuppressants such as cyclosporin A or azathioprine within 6 weeks prior to the screening
* Serious life-threatening conditions
* Allergies to anesthesia
* Subject who is pregnant or nursing
* Subject is on chronic immunosuppressive transplant therapy
* Subjects who tested positive for HIV 1/2, HBV, HCV, HTLV I/II, WNV, and syphilis
* Flu symptoms
* Any past history of lipid disorders: lipedema, lipomatosis, or lipodystrophies
* Active cancer, chemotherapy, or other malignancies in the last 6 months prior to the screening
* Any past history of DVT or pulmonary embolism requiring anticoagulants or other medicines
* Requiring supplemental oxygen
* Major surgeries within 6 months prior to the screening
* Wounds/sepsis ongoing or within 3 months prior to the screening
* Any illness which in the Investigator's judgment, may interfere with the subject's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) Occurring in Less Than 5% of Participants | 30 months
Change from Baseline in Insulin Requirements at 6 Months Post-Treatment | 30 months

SECONDARY OUTCOMES:
Change from Baseline in Glucagon-Stimulated C-Peptide Levels at 6 Months Post-Treatment | 30 months
Change from Baseline in HbA1c Levels | 30 months